CLINICAL TRIAL: NCT04030208
Title: Evaluating Safety and Efficacy of Umbulizer in Patients Requiring Intermittent Positive Pressure Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umbulizer LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1
Record Dates: First submitted 2019-07-09; First posted 2019-07-23 (Actual); Last update posted 2020-08-06 (Actual); Status verified 2020-08

CONDITIONS: Respiratory Failure; Respiratory Insufficiency; Respiratory Arrest
Keywords: respiratory disease; low resource settings; mechanical ventilation; ventilator performance; comparative study; patient safety; ease of use
MeSH Terms: conditions — Respiratory Insufficiency; Apnea; Respiration Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence A (Other): If patient is randomly assigned to Sequence A, they will be placed on a traditional ventilator for the first period. This period will be 1 hour in duration. Delivered tidal volume, respiratory rate (RR), and peak pressure will be recorded throughout the period using the ventilator. Heart rate (HR), Blood Pressure (BP), and oxygen (O2) saturation measurements will be recorded every 5 minutes. Arterial blood gas (ABG) data will be taken at t = 1 hour if the patient is stable on the traditional ventilator. ABGs may be taken more frequently if the patient is destabilizing. Next, the study participant will be transitioned to the Umbulizer to begin Period 2. This period will also be 1 hour in duration. Delivered tidal volume, RR, and peak pressure will be recorded throughout the period using Umbulizer. HR, BP, O2 saturation measurements will be taken every 5 minutes. ABG data will be taken at t = 30 minutes and 1 hour.
  Interventions: Device: Umbulizer; Device: Traditional Mechanical Ventilator
- Sequence B (Other): If patient is randomly assigned to Sequence B, they will be shifted to the Umbulizer for the first period. This period will be 1 hour in duration. Delivered tidal volume, RR, and peak pressure will be recorded throughout the period using Umbulizer. HR, BP, O2 saturation measurements will be recorded every 5 minutes. ABG data will be taken at t = 30 minutes and 1 hour. Next, the study participant will be transitioned to a traditional ventilator to begin Period 2. This period will also be 1 hour in duration. Delivered tidal volume, RR, and peak pressure will be recorded throughout the period using the ventilator. HR, BP, O2 saturation measurements will be recorded every 5 minutes. ABG data will be taken at t = 1 hour if the patient is stable on the traditional ventilator. ABGs may be taken more frequently if the patient is destabilizing.
  Interventions: Device: Umbulizer; Device: Traditional Mechanical Ventilator

INTERVENTIONS:
Device: Umbulizer — Umbulizer is a reliable, user-friendly, and portable system that provides consistent air to the patient by quantitatively delivering a pre-determined tidal volume, inhale/exhale (I/E) ratio, peak pressure, and breathing rate (BPM). It can be configured to deliver either controlled ventilation or assist-controlled ventilation.
Device: Traditional Mechanical Ventilator — A medical device designed to artificially perform breathing functions for patients who are unable to adequately perform these functions on their own.

SUMMARY:
Randomized, control crossover study comparing Umbulizer's efficacy to traditional mechanical ventilators

DETAILED DESCRIPTION:
Mechanical ventilators cost tens of thousands of dollars, rendering them difficult for low and middle income countries to procure. Given chronic shortages of these devices in places like Pakistan, patients are often ventilated manually with Ambu Bags for hours or days. This method is not suitable for long term ventilation and is extremely life threatening.

Umbulizer seeks to reduce preventable deaths due to ventilator scarcity by providing a reliable alternative. The device is accurate, low-cost, and portable, and is an ideal solution for treating patients with respiratory diseases in low-resource settings. The primary objective of this study is to test efficacy and determine non-inferiority of this device in comparison to ventilation provided by traditional ventilators. Secondary objectives of this study include:

1. Testing safety of the device for use over a predetermined period of time
2. Evaluating patient comfort during ventilation with this device
3. Assessing ease of use of this device for doctors and medical staff

ELIGIBILITY:
Inclusion Criteria:

1) Patients needing mechanical ventilation

Exclusion Criteria:

1. Patients with significant airway resistance (i.e. severe chronic obstructive pulmonary disease or asthma) where clinical investigator is concerned about gas trapping or barotrauma
2. Patients with very low lung compliance (i.e. severe acute respiratory distress syndrome or restrictive disease) where clinical investigator is concerned about problems delivering sufficient tidal volume or end expiratory pressure
3. Patients who experienced a myocardial infarction within the last 6 weeks
4. Patients who are determined by a clinical investigator to be too hemodynamically unstable to be enrolled

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-09-04 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Partial Pressure of Carbon Dioxide (PaCO2) | 2 hours
  PaCO2 in mmHg at t = 1 hr (from Arterial Blood Gas or ABG readings) when patient is on Umbulizer compared to PaCO2 at t = 1 hr when patient is on a traditional mechanical ventilator
pH | 2 hours
  pH at t = 1 hr (from ABG readings) when patient is on Umbulizer compared to pH at t = 1 hr when patient is on a traditional mechanical ventilator

SECONDARY OUTCOMES:
Number of Adverse Events | 2 hours
  Number of adverse events on Umbulizer compared to on a traditional ventilator

OTHER OUTCOMES:
Level of Comfort | 2 hours
  Level of comfort on Umbulizer will be determined based on a 4-point scale assessing a combination of indicators (1 point will be assigned for the absence of each of the following: substantial deviation of heart rate from baseline, substantial deviation of blood pressure from baseline, grimacing, diaphoresis).
Ease of Use | 2 hours
  Umbulizer's ease of use will be determined based on survey responses by doctors/medical staff at the end of each experiment
Partial Pressure of Oxygen (PaO2) | 2 hours
  PaO2 in mmHg at t = 1 hr (from ABG readings) when patient is on Umbulizer compared to PaO2 at t = 1 hr when patient is on a traditional mechanical ventilator
O2 Saturation | 2 hours
  O2 saturation (from pulse oximeter) when patient is on Umbulizer compared to when patient is on a traditional mechanical ventilator

CONTACTS AND LOCATIONS:
Overall Officials: Kamran Chima, MBBS, Principal Investigator — Services Hospital
Locations (1):
- Services Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided